CLINICAL TRIAL: NCT01154517
Title: Utility of the History and Physical Exam in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Responsible Party: Peter Lunny, Henry Ford
Other Study IDs: 3617
Record Dates: First submitted 2010-06-30; First posted 2010-07-01 (Estimated); Last update posted 2010-07-01 (Estimated); Status verified 2009-07

CONDITIONS: Abdominal Pain; Back Pain; Dyspnea; Headache; Weakness
MeSH Terms: conditions — Abdominal Pain; Back Pain; Dyspnea; Headache; Asthenia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study is trying to prove that the history and physical exam (H&P) in the emergency department is the most important tool in exam of patients. The investigator is attempting to correlate the time of the H&P of residents and attendings to the accuracy of diagnosis.

DETAILED DESCRIPTION:
The purpose of the study is to examine the utility of the history and physical exam in the emergency room towards obtaining a diagnosis. The goal of this observational study is to correlate physician level of experience and time spent on history and physical exam, to the correct diagnosis.

The aim of this study is:

1. To draw a connection between time and accuracy of the history and physical exam.
2. To draw a connection between time and level of experience as a physician based on post-graduate level.
3. To assess the number of laboratory and radiographic studies and the post-graduate level.
4. To assess the relevance of the labs and radiographs ordered. (Relevance is defined as something that changes plan of care.)

Time is a critical component of the ED physician. Our study will analyse if modern medicine has created a more laboratory/image based need to ascertain a diagnosis or if history and physical examination alone can predict the ultimate diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Anyone over the age of 18 with a generalized complaints able to provide consent

Exclusion Criteria:

* Anyone under 18 yrs and anyone with a very specific, system based complaint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Emergency Department Patients
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2009-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Stevenson, DO, Study Director — Henry Ford Macomb
Locations (1):
- Henry Ford Macomb Hospital, Clinton Township, Michigan, United States